CLINICAL TRIAL: NCT00442286
Title: Rheos® Pivotal Trial: Rheos™ Baroreflex Hypertension Therapy System
Brief Title: Rheos® Pivotal Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 360009
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure; Blood Pressure; Cardiovascular Disease; Resistant Hypertension; Stage 2 Hypertension; Hypertension that is resistant to treatment
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- On (Experimental): Subject will be randomized to a 2:1 allocation to the Rheos ON or OFF arms at the time of Rheos System activation (time point 0). After the six month follow up evaluation, all subjects will have therapy activated, though subjects and treating physicians will not be informed of randomized treatment assignment.
  Interventions: Device: Rheos® Baroreflex Hypertension System
- Off (Experimental): Subject will be randomized to a 2:1 allocation to the Rheos ON or OFF arms at the time of Rheos System activation (time point 0). After the six month follow up evaluation, all subjects will have therapy activated, though subjects and treating physicians will not be informed of randomized treatment assignment.
  Interventions: Device: Rheos® Baroreflex Hypertension System

INTERVENTIONS:
Device: Rheos® Baroreflex Hypertension System — Electrical activation of the Carotid Baroreflex

SUMMARY:
The purpose of this clinical trial is to demonstrate the efficacy and safety of the Rheos system in subjects with hypertension that are resistant to treatment with at least three anti-hypertension agents, one of which is a diuretic.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age and no more than 80 years of age.
* Have been assessed with bilateral carotid bifurcations that are easily interrogated by carotid duplex ultrasound and are below the level of the mandible.
* Office cuff systolic blood pressure greater than or equal to 160 mmHg and have a diastolic blood pressure greater than or equal to 80 mmHg as well as a 24-hour ambulatory systolic blood pressure greater than or equal to 135 mmHg despite at lest one month of maximally tolerated therapy with at least three anti-hypertensive medications, of which at least one must be a diuretic.
* Must have completed the drug compliance questionnaire and have been judged to be compliant with medications.
* For subjects that have had prior bariatric surgery, they must be at least 1 year post-surgery and at a stable weight.
* If female, the subject must be surgically sterile, or using a medically accepted method of birth control and agree to continue use of this method for the duration of the trial. Women of childbearing potential must have a negative serum pregnancy test in the pre-implant blood evaluation.
* Must be an appropriate or reasonable surgical candidate.
* Have signed a CVRx approved informed consent form for participation in this study

Exclusion Criteria:

* Have known or suspected baroreflex failure or autonomic neuropathy.
* Have an arm circumference greater than 46 cm and/or body mass index of greater than 45.
* Have significant cardiac bradyarrhythmias.
* Have chronic atrial fibrillation.
* Have significant orthostatic hypotension
* Had a solid organ or hematologic transplant.
* Had a myocardial infarction, unstable angina, syncope, or cerebral vascular accident within the past 3 months.
* Have carotid atherosclerosis producing a 50% or greater reduction in linear diameter as determined by ultrasound or angiographic evaluation as determined within 6 months of enrollment in the trial.
* Have ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation.
* Have prior surgery, radiation, or endovascular stent placement in either carotid sinus region.
* Have severe chronic kidney disease as defined by:

  * Currently undergoing dialysis or dialysis is planned within 3 months of the implant date
  * eGFR of ≤30 ml/min/1.73m²
* Have hypertension secondary to an identifiable and treatable cause other than sleep apnea.
* Have clinically significant cardiac structural valvular disease.
* Have clinically significant reactive airway disease, chronic obstructive pulmonary disease, and/or primary pulmonary hypertension.
* Have an uncontrolled comorbid medical condition that would adversely affect participation in the trial.
* Have a clinically significant psychological illness that would prohibit the subject's ability to meet the protocol requirements
* Are currently taking an imidazolone receptor agonist
* Are unable or unwilling to fulfill the protocol medication compliance and follow-up requirements.
* Have an active infection within the last month.
* Have a co-morbid condition that reduces life expectancy to less than one year.
* Are enrolled in another concurrent clinical trial, without prior approval of CVRx.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2006-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sanchez, MD, Principal Investigator — Washington University School of Medicine; Mitra Nadim, MD, Principal Investigator — University of Southern California
Locations (44):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Apex Cardiology, Inglewood, California
  - University of Southern California, Los Angeles, California
  - St Joseph Health, Orange, California
  - George Washington University Hospital, Washington D.C., District of Columbia
  - VA Medical Center, Washington D.C., District of Columbia
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Florida Hospital Cardiovascular Institute, Orlando, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - The Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Florida Cardiovascular Institute, Tampa, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - University of Chicago, Dept. of Medicine, Section of Endocinology, Diabetes & Metabolism, Chicago, Illinois
  - The Care Group, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - The Center for Cardiovascular Studies, LLC, Shawnee Mission, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Rex HealthCare, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State Medical Center, Columbus, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Temple University Health System, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Sanford Clinical Research, Sioux Falls, South Dakota
  - Clinical Research Solutions, P.C., Knoxville, Tennessee
  - Saint Thomas Research Institute, Nashville, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas
  - Scott and White Memoral Hospital, Temple, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- Medizinische Hochschule Hannover, Hanover, Germany
- University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Wachter R, Halbach M, Bakris GL, Bisognano JD, Haller H, Beige J, Kroon AA, Nadim MK, Lovett EG, Schafer JE, de Leeuw PW. An exploratory propensity score matched comparison of second-generation and first-generation baroreflex activation therapy systems. J Am Soc Hypertens. 2017 Feb;11(2):81-91. doi: 10.1016/j.jash.2016.12.003. Epub 2016 Dec 16. PMID 28065708
- [Derived] de Leeuw PW, Alnima T, Lovett E, Sica D, Bisognano J, Haller H, Kroon AA. Bilateral or unilateral stimulation for baroreflex activation therapy. Hypertension. 2015 Jan;65(1):187-92. doi: 10.1161/HYPERTENSIONAHA.114.04492. Epub 2014 Oct 20. PMID 25331845
- See also: Additional information about the Rheos Pivotal Trial for patients and medical professionals can be found at http://www.bloodpressuretrial.com/ — http://www.bloodpressuretrial.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 591 patients enrolled, 78 withdrew prior to implant and 187 screen-failed. 4 implants were unsuccessful, and 2 randomized patients were terminated prior to the randomization visit. 55 patients were roll-in patients that were not randomized. A total of 265 patients were both randomized and implanted.
Groups:
- Rheos® Device On; Rheos® Device Off: Subject will be randomized to a 2:1 allocation to the Rheos ON or OFF arms at the time of Rheos System activation (time point 0). After the six month follow up evaluation, all subjects will have therapy activated, though subjects and treating physicians will not be informed of randomized treatment assignment.
  Rheos® Baroreflex Hypertension System: Electrical activation of the Carotid Baroreflex
Period: Overall Study
Arm/Group | Rheos® Device On | Rheos® Device Off
Started | 181 | 84
6 Months | 177 | 83
12 Months | 174 | 82
Completed | 174 | 82
Not Completed | 7 | 2
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — System explanted | 1 | 0
Not completed — Patient Injury | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Roll-In: Subjects that were not included in endpoint analyses
- Total: Total of all reporting groups
Arm/Group | Roll-In | Rheos® Device On | Rheos® Device Off | Total
Number analyzed (Participants) | 55 | 181 | 84 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 151 | 75 | 272
  >=65 years | 9 | 30 | 9 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 65 | 38 | 127
  Male | 31 | 116 | 46 | 193
Race/Ethnicity, Customized [Number; unit: Participants]
  African American | 11 | 30 | 18 | 59
  Hispanic | 3 | 2 | 4 | 9
  White/Caucasian | 40 | 146 | 59 | 245
  Other | 1 | 3 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 | 8 | 5 | 13
  United States | 55 | 165 | 74 | 294
  Germany | 0 | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With a 10mmHg or Greater Reduction in Office Cuff Systolic Blood Pressure
Description: Compare Group A (Rheos® Device On ) versus Group B (Rheos® Device Off) via a double-blind, randomized, parallel group, super-superiority design for proportion of subjects that achieve at least a 10 mm Hg drop in systolic blood pressure at Month 6 compared to Month 0, with a superiority margin of 20%.
Time Frame: 6 months post-activation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheos® Device On | Rheos® Device Off
Number analyzed (Participants) | 181 | 84
percentage of participants | 54.1 [46.9 to 61.4] | 46.4 [35.8 to 57.1]

2. Primary Outcome: Percent of Group A (Rheos® Device On) Patients Who Maintain a 10 mm Hg Drop in Systolic Blood Pressure at 12 Months Post-activation, and Whose Response at 12 Months is at Least 50% of the Response Observed at 6 Months Post-activation.
Description: Compare the sustained response in SBP Month 12 in Group A ( Rheos® Device On ) responders at Month 6 to an objective performance criterion of 65%. A sustained response to therapy required the reduction from Month 0 to Month 12 to be at least 10 mmHg and to remain at least 50% of that seen at Month 6.
Time Frame: 12 months post-activation
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Rheos® Device On
Number analyzed (Participants) | 97
percentage of participants | 87.6 [81.1 to NA] — Lower one-sided 97.5% confident bound interval was used

3. Primary Outcome: Serious Procedure- or System-related Adverse Event-free Rate in Both Implanted and Attempted Patients
Description: Compare the serious procedure- or system-related adverse event-free rate for events occurring within 30 days of implant to a pre-specified objective performance criterion of 82% set based on historical literature on implantable cardioverter defibrillators (ICD) and pacemakers.
  Note: The purpose of this outcome measure was to evaluate the effect of having the device implanted, not to compare the outcomes between the two treatment groups. Therefore, both groups were analyzed as a single cohort.
Time Frame: 30 days post implant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Implanted or Attempted Patients: All Implanted or Attempted patients enrolled in the study. Roll-ins were excluded.
Arm/Group | All Implanted or Attempted Patients
Number analyzed (Participants) | 270
percentage of participants | 74.8 [70.5 to NA] — Lower one-sided 95% confidence bound interval was used

4. Primary Outcome: Major Hypertension-related and Serious Device-related Adverse Event-Free Rate in Both Implanted and Attempted Patients.
Description: Compare the event-free rate for all major hypertension-related and serious device-related adverse events occurring between 30 days post-implant and the Month 12 visit, to a pre-specified objective performance criterion of 72% based on similar implantable devices such as defibrillators and resynchronization devices.
  Note: The purpose of this outcome measure was to evaluate the effect of having the device implanted, not to compare the outcomes between the two treatment groups. Therefore, both groups were analyzed as a single cohort.
Time Frame: 12 months-post activation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Implanted or Attempted Patients: All Implanted or Attempted patients active at 30 days post-implant. Excludes roll-in patients.
Arm/Group | All Implanted or Attempted Patients
Number analyzed (Participants) | 266
percentage of participants | 87.2 [83.8 to NA] — Lower One-sided 95% confident bound interval was used.

5. Primary Outcome: Therapy-related Adverse Event-free Rate.
Description: Compare Group A (Rheos® Device On ) versus Group B (Rheos® Device Off) therapy-related adverse event-free rates via a double-blind, randomized, parallel group, non-inferiority design for therapy-related serious adverse events occurring between 30 days post-implant and the Month 6 visit. The non-inferiority margin was 15%.
Time Frame: 6 months post-activation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheos® Device On | Rheos® Device Off
Number analyzed (Participants) | 181 | 84
percentage of participants | 91.7 [87.7 to 95.7] | 89.3 [82.7 to 95.9]

ADVERSE EVENTS:
Time Frame: 12 months post-randomization
Description: Due to the learning curve associated with the implant of the Rheos system, the initial subjects (up to a maximum of two) at each center that had not been previously implanted with the Rheos system will be non-randomized roll-in subjects. These subjects were not subjected to the formal efficacy and safety analysis process.
Arm/Group | Rheos® Device On | Rheos® Device Off
Serious Adverse Events (participants affected / at risk) | 102/181 | 45/84
Other Adverse Events (participants affected / at risk) | 75/181 | 39/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheos® Device On (N=181) | Rheos® Device Off (N=84)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Congestive cardiac failure (Cardiac disorders) | 4 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischemia (Cardiac disorders) | 1 | 0
Unstable Angina (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 0
Miosis (Eye disorders) | 1 | 0
Retinitis (Eye disorders) | 1 | 0
Unilateral Blindness (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Ischemic Colitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 1 | 0
Ulcerative Colitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 11 | 3
Death (General disorders) | 1 | 1
Implant site pain (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Edema (General disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Neck Abscess (Infections and infestations) | 1 | 0
Anogenital warts (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Viral Meningitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Device lead damage (Injury, poisoning and procedural complications) | 2 | 0
Device migration (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Incision site infection (Injury, poisoning and procedural complications) | 0 | 1
Medical device pain (Injury, poisoning and procedural complications) | 2 | 1
Nerve injury (Injury, poisoning and procedural complications) | 6 | 3
Open wound (Injury, poisoning and procedural complications) | 0 | 1
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound infection (Injury, poisoning and procedural complications) | 1 | 0
XIIth nerve injury (Injury, poisoning and procedural complications) | 3 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 3
Diplegia (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 1 | 3
Thalamus hemorrhage (Nervous system disorders) | 1 | 0
Tongue paralysis (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Psychiaric symptom (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 1 | 0
Chronic renal failure (Renal and urinary disorders) | 0 | 1
Renal artery fibromusular dysplasia (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Face swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial Bypass Operation (Surgical and medical procedures) | 1 | 0
Cyst removal (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Malignant tumor excision (Surgical and medical procedures) | 0 | 1
Mass excision (Surgical and medical procedures) | 0 | 1
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Accelerated Hypertension (Vascular disorders) | 2 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 0
Hemotoma (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 5 | 1
Hypertensive crisis (Vascular disorders) | 10 | 8
Hypertensive emergency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 6 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rheos® Device On (N=181) | Rheos® Device Off (N=84)
Chest Pain (General disorders) | 11 | 1
Fatique (General disorders) | 8 | 6
Local swelling (General disorders) | 2 | 5
Pheripheral edema (General disorders) | 4 | 5
Nasopharyngitis (Infections and infestations) | 5 | 5
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 10 | 4
Gout (Metabolism and nutrition disorders) | 2 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 11 | 3
Dizziness (Nervous system disorders) | 6 | 6
Headache (Nervous system disorders) | 24 | 5
Hypoaesthesia (Nervous system disorders) | 17 | 4
Hypotension (Vascular disorders) | 19 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site must notify CVRx and a designated Publication Committee 30 days before submission. The complete text of the publication is required for review. If CVRx does not respond within 30 days of the date received by CVRx, the site may proceed with publication. If CVRx determines that there are changes to be made, the publication maybe delayed for up to 90 days. The site must not submit a publication without the satisfaction of the Publication Committee.